CLINICAL TRIAL: NCT07352878
Title: Evaluation of the Quality of Life in Patients With Chronic Iron Overload Due to Hemoglobinopathies in Greece, Who Are Under Treatment With Deferasirox, Based on Standard Clinical Practice.
Brief Title: Evaluation of the Quality of Life in Patients With Chronic Iron Overload Due to Hemoglobinopathies in Greece.
Acronym: FEROUSA
Status: Not yet recruiting | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Collaborators: Aghia Sophia Children's Hospital of Athens (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-DEF-EL-256
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Thalassemia; Iron Overload
Keywords: quality of life; iron overload; treatment satisfaction
MeSH Terms: conditions — Thalassemia; Iron Overload

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational clinical study aims to evaluate the HRQoL of thalassemia patients with iron overload in Greece, who are under treatment with deferasirox based on standard clinical practice.

DETAILED DESCRIPTION:
The assessment of health-related quality of life (HRQoL) in thalassemic patients with iron overload offers a holistic approach to the disease and leads to better communication between physicians and patients. This prospective, non-interventional, observational clinical study aims to evaluate the HRQoL, adherence to deferasirox treatment and treatment effectiveness as well as patients' satisfaction and safety with deferasirox.

All participants will complete a set of questionnaires and scales for QoL, adherence to treatment, and satisfaction of the treatment for iron overload. Demographic and clinical characteristics will be recorded to define patient subgroups based on the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult patients (≥ 18 years). 2. Patients with major beta-thalassemia with iron overload due to frequent blood transfusions (≥7 ml/kg/month of packed red blood cells).

  3. Patients with chronic iron overload due to blood transfusions if deferoxamine therapy is contraindicated or insufficient in the following patient groups:
  * adult patients with major beta-thalassemia with iron overload due to infrequent blood transfusions (<7 ml/kg/month of packed red blood cells).
  * adult patients with other types of anemia.

    4. Patients with non-transfusion-dependent thalassemia syndromes with chronic iron overload requiring chelation therapy when deferoxamine therapy is contraindicated or insufficient.

    5. Patients who were receiving deferasirox before their inclusion in the study (90, 180, 360, 900 mg) and at their inclusion require treatment with deferasirox at least 900 mg, as part of the treatment of chronic iron overload and according to the SPC.

    6. Consent and compliance of participants with the treatments and procedures of the study.

    7. Patients for whom data from the last six months from the date of inclusion (medical history, concomitant medication) are available to determine the endpoints.

Exclusion Criteria:

* 1. Patients under 18 years of age. 2. Patients with myelodysplastic syndromes. 3. Patients with a contraindication to taking deferasirox 90, 180, 360, 900 mg according to the drug's SmPC.

  4. Patients receiving or expect to receive another chelating agent (e.g. deferoxamine, deferiprone) in addition to deferasirox, during the study.

  5. Patients with a history of mental illness, substance abuse, to a degree that may prevent their participation in the study.

  6. Patients are participating in another research protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with major beta-thalassemia with iron overload due to frequent blood transfusions (≥7 ml/kg/month of packed red blood cells) will be included in the study and who were receiving deferasirox before their inclusion in the study (90, 180, 360, 900 mg) and at their inclusion require treatment with deferasirox at least 900 mg, as part of the treatment of chronic iron overload and according to the SPC.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of health-related quality of life in patients with chronic iron overload | Score of the Short-Form 36-item Health Survey (SF-36v2) questionnaire at baseline, at 6 and at 12 months and the change from baseline and among at 6 and 12 months
  Score of the Short-Form 36-item Health Survey (SF-36v2) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Ginis, MD, Study Director — Elpen Pharmaceutical Co. Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kattamis A, Aydinok Y, Taher A. Optimising management of deferasirox therapy for patients with transfusion-dependent thalassaemia and lower-risk myelodysplastic syndromes. Eur J Haematol. 2018 Sep;101(3):272-282. doi: 10.1111/ejh.13111. Epub 2018 Jul 27. PMID 29904950
- [Background] Voskaridou E, Kattamis A, Fragodimitri C, Kourakli A, Chalkia P, Diamantidis M, Vlachaki E, Drosou M, Lafioniatis S, Maragkos K, Petropoulou F, Eftihiadis E, Economou M, Klironomos E, Koutsouka F, Nestora K, Tzoumari I, Papageorgiou O, Basileiadi A, Lafiatis I, Dimitriadou E, Kalpaka A, Kalkana C, Xanthopoulidis G, Adamopoulos I, Kaiafas P, Mpitzioni A, Goula A, Kontonis I, Alepi C, Anastasiadis A, Papadopoulou M, Maili P, Dionisopoulou D, Tsirka A, Makis A, Kostaridou S, Politou M, Papassotiriou I; Greek Haemoglobinopathies Study Group. National registry of hemoglobinopathies in Greece: updated demographics, current trends in affected births, and causes of mortality. Ann Hematol. 2019 Jan;98(1):55-66. doi: 10.1007/s00277-018-3493-4. Epub 2018 Sep 8. PMID 30196444
- [Background] Arian M, Mirmohammadkhani M, Ghorbani R, Soleimani M. Health-related quality of life (HRQoL) in beta-thalassemia major (beta-TM) patients assessed by 36-item short form health survey (SF-36): a meta-analysis. Qual Life Res. 2019 Feb;28(2):321-334. doi: 10.1007/s11136-018-1986-1. Epub 2018 Sep 7. PMID 30194626
- [Background] Tartaglione I, Origa R, Kattamis A, Pfeilstocker M, Gunes S, Crowe S, Fagan N, Vincenzi B, Ruffo GB. Two-year long safety and efficacy of deferasirox film-coated tablets in patients with thalassemia or lower/intermediate risk MDS: phase 3 results from a subset of patients previously treated with deferasirox in the ECLIPSE study. Exp Hematol Oncol. 2020 Aug 10;9:20. doi: 10.1186/s40164-020-00174-2. eCollection 2020. PMID 32793403
- [Background] Goulas V, Kouraklis-Symeonidis A, Manousou K, Lazaris V, Pairas G, Katsaouni P, Verigou E, Labropoulou V, Pesli V, Kaiafas P, Papageorgiou U, Symeonidis A. A multicenter cross-sectional study of the quality of life and iron chelation treatment satisfaction of patients with transfusion-dependent beta-thalassemia, in routine care settings in Western Greece. Qual Life Res. 2021 Feb;30(2):467-477. doi: 10.1007/s11136-020-02634-y. Epub 2020 Sep 13. PMID 32920766
- [Background] Lai YR, Cappellini MD, Aydinok Y, Porter J, Karakas Z, Viprakasit V, Siritanaratkul N, Kattamis A, Liu R, Izquierdo M, Lasher J, Govindaraju S, Taher A. An open-label, multicenter, efficacy, and safety study of deferasirox in iron-overloaded patients with non-transfusion-dependent thalassemia (THETIS): 5-year results. Am J Hematol. 2022 Aug;97(8):E281-E284. doi: 10.1002/ajh.26592. Epub 2022 May 27. No abstract available. PMID 35560253
- [Background] Klonizakis P, Klaassen R, Sousos N, Liakos A, Tsapas A, Vlachaki E. Evaluation of the Greek TranQol: a novel questionnaire for measuring quality of life in transfusion-dependent thalassemia patients. Ann Hematol. 2017 Nov;96(11):1937-1944. doi: 10.1007/s00277-017-3122-7. Epub 2017 Sep 7. PMID 28884221